CLINICAL TRIAL: NCT02660593
Title: SanGrow Decoction in Patients With Diabetes- Single Center, Open, and Non-randomized Study
Brief Title: Efficacy and Safety ofSanGrow Decoction for Patients With Diabetes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shidaihuajing Institute for Diabetic Research (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SanGrow Decoction for diabetes
Record Dates: First submitted 2016-01-17; First posted 2016-01-21 (Estimated); Last update posted 2016-04-27 (Estimated); Status verified 2016-01

CONDITIONS: Diabetes Mellitus
Keywords: Diabetes Mellitus; Chinese medicine; exercise; diet
MeSH Terms: conditions — Diabetes Mellitus; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SanGrow (Experimental): Patients will be given SanGrow Decoction 150 ml per day for 3 months.
  Interventions: Dietary Supplement: SanGrow Decoction

INTERVENTIONS:
Dietary Supplement: SanGrow Decoction — SanGrow Decoction is perpared according to the principle of Chinese medicine to treat thirsty and maransis.

SUMMARY:
MedlinePlus related topics: Blood Sugar

Primary Outcome Measures:

* Fast glucose and HbA1c change between the baseline and end of study [ Time Frame: From baseline to 30 and 100 days]
* [ Designated as safety issue: No ]
* Successful rate of blood glucose control (the proportion of patients with HbA1c <7%) [ Time Frame: From baseline to 30 days and 100 days] [ Designated as safety issue: No ]

Secondary Outcome Measures:

• To evaluate the change of quality of life in the 1 months by the health questionnaire SF-36 [ Time Frame: From baseline to month 1 ] [ Designated as safety issue: No ]

DETAILED DESCRIPTION:
This study is aimed to evaluate the safety and efficacy of Sangrow Decotion, diet and exercise for the treatment of type 2 diabetes. Previous study has shown that this therapeutic regimen is safe and effective.

ELIGIBILITY:
Inclusion Criteria:

* Type II diabetes mellitus patients who have received medical treatment for more than 3 months
* Patients willing to sign written informed consent form

Exclusion Criteria:

* Patients unable or unwilling to comply with the requirements of the protocol
* Females who are pregnant or nursing or females of childbearing potential who are unwilling to maintain contraceptive therapy for the duration of the study
* Life expectancy < 6 months due to concomitant illnesses.

Ages: 10 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-03; Primary Completion 2017-03 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Blood Sugar level | From baseline to 30 and 90 days
  Fast glucose change between the baseline and end of study

CONTACTS AND LOCATIONS:
Overall Officials: Shizhan CHi, PhD, Study Chair — Shidaihuajing Institute
Locations (2):
- China (2):
  - Jiuhua Hospital, Beijing, Beijing Municipality
  - Xuanwu Hospital, Beijing, Beijing Municipality

IPD SHARING:
Plan to Share IPD: No